CLINICAL TRIAL: NCT02780531
Title: Genetic and Blood Biomarkers in Subjects With Neurological and Neuromuscular Diseases
Brief Title: Genetic and Blood Biomarkers in Neurological and Neuromuscular Diseases
Acronym: Neurogenetic
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jafar Kafaie, MD, Assistant Professor, St. Louis University
Other Study IDs: 25726
Record Dates: First submitted 2016-04-07; First posted 2016-05-23 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Neurological Disorders; Neuromuscular Disorders
MeSH Terms: conditions — Nervous System Diseases; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood: Blood is the preferred sample to be collected as it yields the broadest number of components to be studied, including deoxyribonucleic acid ("DNA"), ribonucleic acid ("RNA"), protein & lymphocytes (approximately 10 milliliters). These may be immediately utilized or frozen -80C for future research.
  Other tissues: In some circumstances, a subject may have undergone or will undergo a clinical procedure yielding bodily tissues or fluids (e.g. a muscle, tumor biopsy, spinal tap). If this is the case, nucleic acids (DNA & RNA) and proteins can be extracted for study. Furthermore, there may be rare cases where comparisons between blood DNA & tissue DNA/RNA is needed (e.g. a mutation identified is predicted to affected splicing which can only be verified by studying the RNA from tissues).
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify genetic or other factors in the subjects blood that may predispose them to getting a particular disease or tell researchers how the disease will behave, for example how fast it will progress or what areas of the body might be affected. A second goal is to relate such factors to how such a condition affects the subjects clinically as well as how it affects the electrical functions of nerves and muscles.

DETAILED DESCRIPTION:
The etiology of many neurological and neuromuscular disorders is largely unknown. Contributions likely come from both inherited and environmental factors. Amyotrophic lateral sclerosis ("ALS") is a prototypical example. In 5-10% of cases, genetic mutations exert a strong enough influence on disease development that the syndrome is transmitted in a clearly Mendelian fashion. Investigations in these "familial" ALS cases have identified more than 20 causative disease genes. Intensive study of these genes has helped identify several key cellular pathways as important for disease, not only in cases with obvious gene mutations, but even in the 90% of ALS cases that appear to be "sporadic." Further insights have come from investigating blood biomarkers in ALS such as gene and protein expression and lymphocyte profiling. It is hoped that further genetic and biomarker analysis will identify additional genetic risk factors or biomarkers to better understand the disease and improve therapeutic development. These advances can be applied not just to ALS but to the broad range of neurological and neuromuscular diseases, including Charcot Marie Tooth neuropathy, the muscular dystrophies, epilepsies, Parkinson's disease, and Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be individuals with neurologic or neuromuscular disease who are deemed well-enough for sample collection.

Exclusion Criteria:

* Subjects who are not willing to undergo sample collection, genetic analysis, or unwilling to share clinical information or their samples.
* Pregnant women will also be excluded.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 350 study subjects per year will be recruited from neurology and neuromuscular clinics and inpatient services of St. Louis University and Cardinal Glennon Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Recognizing possible pathogenic mutation in specific genes | 2 years
  Genetic test by collection of blood including whole exome sequencing and targeted gene sequencing

SECONDARY OUTCOMES:
Abnormal protein and enzyme structure and function that may explain a particular disease or syndrome | 2 years
  Using epidermal nerve fiber density testing in skin biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Sean Goretzke, MD, Study Chair — St. Louis University
Locations (1):
- Saint Louis University Department of Neurology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No